CLINICAL TRIAL: NCT02387008
Title: Prospective, Comparative Assessment of Alveolar Bone Augmentation Using Guidor Membrane in the Bound Edentulous Space
Brief Title: Prospective, Comparative Assessment of Alveolar Bone Augmentation Using GUIDOR® Membrane in the Bound Edentulous Space
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was halted prematurely by UNC for low accrual.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-2429
Record Dates: First submitted 2015-02-11; First posted 2015-03-12 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- GUIDOR® membrane with FDBA (Active Comparator): horizontal bone augmentation with synthetic GUIDOR® membrane + FDBA
  Interventions: Device: GUIDOR® membrane with FDBA
- GUIDOR® membrane alone (Active Comparator): horizontal bone augmentation with synthetic GUIDOR® membrane
  Interventions: Device: GUIDOR® membrane
- Bio-Gide® membrane with FDBA (Active Comparator): xenograft BioGide® membrane + FDBA
  Interventions: Device: Bio-Gide® membrane with FDBA

INTERVENTIONS:
Device: GUIDOR® membrane with FDBA — horizontal bone augmentation with synthetic GUIDOR® membrane + FDBA
  Arms: GUIDOR® membrane with FDBA
Device: GUIDOR® membrane — horizontal bone augmentation with synthetic GUIDOR® membrane
  Arms: GUIDOR® membrane alone
Device: Bio-Gide® membrane with FDBA — xenograft BioGide® membrane + FDBA
  Arms: Bio-Gide® membrane with FDBA

SUMMARY:
Purpose: The goal of guided bone augmentation is to provide an alveolar ridge of sufficient dimension to permit dental implant placement. While a wide variety of bone graft and barrier membrane products are commercially available, limited evidence exists supporting the use of one technique over another. The purpose of this study is to radiographically define the dimensional bone changes following horizontal bone augmentation using a synthetic GUIDOR® (Sunstar, Inc.) membrane. Secondary outcome measurements will include the assessment of inflammation, infection, or other wound healing complications.

Participants: A total of 60 patients requiring bone augmentation of a single bound edentulous site prior to dental implant placement will be selected for this study. This is a multicenter study with 30 patients receiving treatment at each study site.

Procedures (methods): Patients will be randomly allocated to receive horizontal bone augmentation with synthetic GUIDOR® membrane + freeze dried bone augmentation (FDBA), synthetic GUIDOR® membrane alone, or xenograft BioGide® membrane + FDBA. Cone beam computed tomography (CBCT) imaging will be obtained at baseline and 6 months post-operatively to assess dimensional alveolar ridge changes. Additionally, post-operative appointments at 1, 2, and 4 weeks post-grafting will be completed to assess the presence of inflammation, infection, wound dehiscence, or membrane exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. ≥ 21 years and ≤ 75 years
3. In need of one or more implants replacing missing or non-restorable teeth in the maxilla within region 14 to 24 or the mandible within region 34 to 44
4. Edentulous for at least 6 months at study site
5. A buccal-lingual ridge width at study site of ≤ 4 mm
6. A mesial-distal distance between adjacent teeth at study site at bone level of at least 5 mm
7. A keratinized mid-buccal mucosal thickness of at least 2 mm at study site (measured buccally at MD midline from the mucogingival junction to the projected alveolar ridge crest)
8. Teeth adjacent (mesial and distal) to study site must consist of two stable, natural teeth without signs of periodontal bone loss (> 3 mm) and/or significant soft tissue loss
9. A minimum of twenty teeth in good repair

Exclusion Criteria:

1. Insufficient interocclusal distance for implant placement and restoration at study site
2. More than 3 mm vertical bone loss at study site as measured from the mid-buccal crest of bone on the adjacent teeth
3. Previous site development (soft and/or bone tissue) performed at the study site
4. Untreated rampant caries and uncontrolled periodontal disease
5. A history within the last 6 months of the daily use of any non-cigarette tobacco products (smokeless chewing tobacco, e-cigarette, pipe or cigar smoking), or of smoking more than 10 cigarettes per day.
6. Current alcohol dependency, alcohol abuse or chemical dependency based on DSM-IV Criteria or drug abuse
7. Subjects having uncontrolled endocrine-induced diseases (e.g. uncontrolled diabetes mellitus)
8. Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
9. Use of any substance or medication that will influence bone metabolism (e.g. intravenous bisphosphonates)
10. Need for systemic corticosteroids or any other medication that would influence post-operative healing and/or osseointegration
11. History of radiation in the head and neck region
12. Subject is pregnant as reported at time of enrollment
13. Unable or unwilling to return for follow-up visits for a period of 6 months
14. Unlikely to be able to comply with study procedures according to Investigators judgement
15. Previous enrollment or randomization of treatment in the present study
16. Involvement in the planning/conduct of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cook, DDS MS, Principal Investigator — UNC School of Dentistry
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - University of North Carolina School of Dentistry, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bio-Gide® Membrane With FDBA: Xenograft BioGide® membrane + Freeze-dried Bone Allograft (FDBA)
  Bio-Gide® membrane with FDBA: xenograft BioGide® membrane + FDBA
Period: Overall Study
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
Started | 2 | 0 | 4
Completed | 2 | 0 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the GUIDOR® Membrane Alone Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA | Total
Number analyzed (Participants) | 2 | 0 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 1 |  | 1 | 2
  >=65 years | 1 |  | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2 | 4
  Male | 0 |  | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  | 2 | 4
  Not Hispanic or Latino | 0 |  | 2 | 2
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 2 |  | 4 | 6
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 |  | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dimensional Bone Changes at 6 Months
Description: Dimensional bone changes will assessed by calculating horizontal width and vertical height changes using data from DICOM images acquired by Cone beam computed tomography (CBCT).
Time Frame: 6 months after treatment
Population: Protocol-defined collection intervals were not achieved for any subjects enrolled; therefore, no data available for this measure.
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Inflammation
Description: The presence or absence of soft tissue erythema within 3 mm from the crestal incision in the edentulous site will be visually assessed at post-operative evaluations.
Time Frame: 7 days, 14 days, 28 days, 6 months
Population: No participants were randomized to the GUIDOR® Membrane Alone Arm
Measure: Count of Participants; unit: Participants
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
Number analyzed (Participants) | 2 | 0 | 4
Participants
  Inflammation Present | 0 | 0 | 0
  Inflammation Absent | 2 | 0 | 4

3. Secondary Outcome: Infection
Description: The presence or absence of infection in the area of ridge augmentation will be assessed through visual evaluation and palpation. The presence of suppuration from the crestal incision or soft tissues adjacent to the localized ridge augmentation will be assessed through visual evaluation. Fluctuance in the area of the augmentation will be assessed through gentle palpation of the surgical site.
Time Frame: 7 days, 14 days, 28 days, 6 months
Population: No participants were randomized to the GUIDOR® Membrane Alone Arm
Measure: Count of Participants; unit: Participants
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
Number analyzed (Participants) | 2 | 0 | 4
Participants
  Infection present | 0 | 0 | 0
  Infection absent | 2 | 0 | 4

4. Secondary Outcome: Membrane Exposure
Description: The presence of membrane exposure or soft tissue dehiscence will be visually assessed.
Time Frame: 7 days, 14 days, 28 days, 6 months
Population: No participants were randomized to the GUIDOR® Membrane Alone Arm
Measure: Count of Participants; unit: Participants
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
Number analyzed (Participants) | 2 | 0 | 4
Participants
  membrane exposure or soft tissue dehiscencePresent | 0 | 0 | 0
  membrane exposure or soft tissue dehiscence Absent | 2 | 0 | 4

ADVERSE EVENTS:
Time Frame: From baseline to the completion of trial, approximately 6 months.
Description: No participants were randomized to the GUIDOR® Membrane Alone Arm
Arm/Group | GUIDOR® Membrane With FDBA | GUIDOR® Membrane Alone | Bio-Gide® Membrane With FDBA
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
Slow progression of recruitment and consequent enrollment of only 6 out of 60 planned participants lead to study termination and insufficient data to provide a substantive analysis. Thus data analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02387008/Prot_SAP_000.pdf